CLINICAL TRIAL: NCT06717516
Title: Renal Involvement in Adult Patients with Inflammatory Bowel Disease and Its Relation to Duration and Disease Activity .
Brief Title: Renal Involvement in Adult Patients with Inflammatory Bowel Disease and Its Relation to Duration and Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Abdel-Aal Khalifa Abdel-Aal, Renal Involvement in Adult patients with Inflammatory bowel disease and its relation to duration and disease activity ., Assiut University
Other Study IDs: Renal inolvement in adult IBD
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: IBD and Renal Involement; IBD Activity and Kidney Affection
Keywords: IBD and kidney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To Assess the pattern of renal injury in patients with inflammatory bowel disease and its relation to the duration and disease activity by Identification and characterization of early renal manifestations (e.g., proteinuria, hematuria, electrolyte imbalances) in IBD patients. and know Correlation between kidney involvement and IBD severity, including flare-ups and complications.

and know Impact of early renal manifestations on long-term renal outcomes, such as progression to CKD or development of AKI.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), comprising ulcerative colitis (UC) and Crohn's disease (CD), is a chronic immunemediated disorder of the gastro-intestinal tract characterized by recurrent inflammation and epithelial injury of the intestine. Extraintestinal manifestations are seen in 6% to 47% of patients diagnosed with IBD. Renal and urinary tract involvement occurs in 4% to 23% of patients with IBD, with renal calculi being the most common form of renal involvement. IBD is associated with a range of renal manifestations, including nephrolithiasis, glomerulonephritis, tubulointerstitial nephritis, and secondary amyloidosis, which can lead to acute or chronic renal insufficiency. Several potential mechanisms might contribute to the higher risk of incident CKD and AKI in patients with IBD. First, in the context of IBD, acute or chronic loss of circulating volume (salt and water depletion) due to persistent inflammation of the intestine and repeated intestinal resection could lead to electrolyte abnormalities followed by acute and chronic loss of kidney function, which may not be always reversible. Second, dysbiosis in patients with IBD is associated with increased production of microbiota-derived uremic toxins and microinflammation, both of which promote the progression of renal diseases. Third, IBD-related alterations in the innate and adaptive immune systems may lead to elevated proinflammatory cytokines, which are particularly implicated in the progression of renal disease. Understanding these associations is crucial for management and monitoring of IBD patients, particularly for those who may develop renal complications, so mitigating impact on kidney function and overall health.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Confirmed diagnosis of IBD either crohns disease or ulcerative colities based on clinical ,endoscopic ,histological and radiological findings . - Patients in any stage of IBD, including remission, active disease, and flare-ups. - Willingness to participate and provide informed consent. - Renal Assessment for participants.

Exclusion Criteria:

- Pre-existing chronic kidney disease (CKD) at any stage. - Known primary kidney diseases unrelated to IBD. - Current use of nephrotoxic medications not related to IBD treatment. - Pregnancy or breastfeeding. - Patients who are unable to comply with study protocols or follow-up assessment - Presence of other significant comorbidities that impact renal function or overall health

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older with Confirmed diagnosis of IBD either crohns disease or ulcerative colities based on clinical ,endoscopic ,histological and radiological findings
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Identification of renal manifestations in IBD patients and Correlation between kidney involvement and IBD severity, including flare-ups and complications and its Impact on long-term renal outcomes, such as progression to CKD or development of AKI | scheduled follow-ups at 3,6,12 months
  Identification and characterization of renal manifestations (e.g., proteinuria, hematuria, electrolyte imbalances) in IBD patients and Correlation between kidney involvement and IBD severity, including flare-ups and complications and Impact of early renal manifestations on long-term renal outcomes, such as progression to CKD or development of AKI

CONTACTS AND LOCATIONS:
Overall Officials: Effat AbdelHady Tony Ahmed, Study Chair; Mohammed Abdelhakim Elmahdy, Study Director

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lian X, Wang Y, Wang S, Peng X, Wang Y, Huang Y, Chen W. Does inflammatory bowel disease promote kidney diseases: a mendelian randomization study with populations of European ancestry. BMC Med Genomics. 2023 Sep 26;16(1):225. doi: 10.1186/s12920-023-01644-2. PMID 37752523
- [Background] Evenepoel P, Poesen R, Meijers B. The gut-kidney axis. Pediatr Nephrol. 2017 Nov;32(11):2005-2014. doi: 10.1007/s00467-016-3527-x. Epub 2016 Nov 15. PMID 27848096
- [Background] Kumar S, Pollok R, Goldsmith D. Renal and Urological Disorders Associated With Inflammatory Bowel Disease. Inflamm Bowel Dis. 2023 Aug 1;29(8):1306-1316. doi: 10.1093/ibd/izac140. PMID 35942657
- [Background] Kellum JA, Romagnani P, Ashuntantang G, Ronco C, Zarbock A, Anders HJ. Acute kidney injury. Nat Rev Dis Primers. 2021 Jul 15;7(1):52. doi: 10.1038/s41572-021-00284-z. PMID 34267223
- [Background] van Hoeve K, Hoffman I. Renal manifestations in inflammatory bowel disease: a systematic review. J Gastroenterol. 2022 Sep;57(9):619-629. doi: 10.1007/s00535-022-01903-6. Epub 2022 Jul 14. PMID 35834005
- [Background] Piovani D, Danese S, Peyrin-Biroulet L, Bonovas S. Environmental, Nutritional, and Socioeconomic Determinants of IBD Incidence: A Global Ecological Study. J Crohns Colitis. 2020 Mar 13;14(3):323-331. doi: 10.1093/ecco-jcc/jjz150. PMID 31504350